CLINICAL TRIAL: NCT03434691
Title: Effects of Dexmedetomidine vs Midazolam on Microcirculation in Septic Shock Patients: a Muscle Microdialysis Study
Brief Title: Effects of Dexmedetomidine vs Midazolam on Microcirculation in Septic Shock Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Military Hospital of Tunis (Other)
Responsible Party: Principal Investigator, Hajjej Zied, Clinical Professor, Military Hospital of Tunis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: DEX03/06
Record Dates: First submitted 2018-02-08; First posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEX group (Experimental): continuous infusion of Dexmedetomidine at 0.4 μg/kg per hour and remifentanyl A microdialysis probe was placed into the femoral quadriceps. An initial set of measurements will be obtained during the sedation with Midazolam and remifentanyl (before randomization). This set of measurements will be considered as baseline. Then samples were collected every 6 hours for 3 days. The changes in the energy-related metabolites lactate, the lactate/pyruvate ratio, glucose and glycerol were analyzed. Concomitantly with dialysate sampling, the effects on global haemodynamics, were assessed. Lactate and L/P clearances were also calculated.
  Interventions: Device: Microdialysis Probe (Muscle microdialysis); Drug: remifentanyl
- MDZ group (Active Comparator): continuous infusion of a Midazolam at 0,1 mg/kg/h and remifentanyl A microdialysis probe was placed into the femoral quadriceps. An initial set of measurements will be obtained during the sedation with Midazolam and remifentanyl (before randomization). This set of measurements will be considered as baseline. Then samples were collected every 6 hours for 3 days. The changes in the energy-related metabolites lactate, the lactate/pyruvate ratio, glucose and glycerol were analyzed. Concomitantly with dialysate sampling, the effects on global haemodynamics, were assessed. Lactate and L/P clearances were also calculated.
  Interventions: Device: Microdialysis Probe (Muscle microdialysis); Drug: remifentanyl

INTERVENTIONS:
Device: Microdialysis Probe (Muscle microdialysis) — Interstitial tissue concentrations of lactate, pyruvate, glucose and glycerol were determined at baseline and then every six hours for the following 72 hours after randomization.
  During the study period, conventional treatment was continued as per usual practice. Fluid challenges were performed, and repeated as necessary, to maintain central venous pressure (CVP) ≥8 and pulmonary arterial occlusion pressure (PAOP) ≥12 mmHg. Norepinephrine was titrated to maintain mean arterial pressure (MAP) ≥65 mmHg. Packed red blood cells were transfused when Hemoglobin (Hb) concentrations decreased below 7 g/dL, or if the patient exhibited clinical signs of inadequate systemic oxygen supply.
Drug: remifentanyl — Only the dose of remifentanyl (initial infusion of 6 µg/kg/h) can be changed to achieve a Goal of sedation: Richmond agitation-sedation scale 0 to -2.

SUMMARY:
To investigate changes in the concentration of glucose, lactate, pyruvate and glycerol in the extracellular fluid of the skeletal muscle following Dexmedetomidine administration in patients with septic shock.

DETAILED DESCRIPTION:
Prospective randomized double blinded study. Investigators planned to enroll 60 cases diagnosed with septic shock All patients will be sedated with Midazolam and remifentanyl in accordance with a local unit protocol.

After a period of six hours of hemodynamic stability, patients were randomized to receive either continuous infusion of Dexmedetomidine at 0.4 μg/kg per hour and remifentanyl (DEX group) or a continuous infusion of a Midazolam and remifentanyl (MDZ Group).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years
* Septic shock requiring norepinephrine (NE) to maintain a mean arterial pressure (MAP) of at least 65mm Hg despite appropriate volume resuscitation (fluid challenge of 20 mL/kg-40 mL/kg)
* Septic shock criteria were defined according to the new Sepsis-3 definition

Exclusion Criteria:

* pregnancy
* uncontrolled hemorrhage
* terminal heart failure
* significant valvular heart disease
* documented or suspected acute coronary syndrome, and limitations on the use of inotropes: left ventricle outflow obstruction, systolic anterior motion of the mitral valve
* refractory bradycardia (heart rate slower than 60 bpm despite of adequate treatment)
* 2nd and 3rd degree of AV-block ,the onset of septic shock more than 24 h before enrollment ,
* APACHE II > 30 at enrollment
* Severe liver cirrhosis (Child B or C)
* New onset of myocardial infarction within 30 days or heart failure (NYHA 4)
* attending other trial in ICU within one month
* allergic history to dexmedetomidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-02-08 (Actual); Primary Completion 2018-11-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
changes in the concentration of glucose(mmol/l) in the extracellular fluid of the skeletal muscle | Time Frame: At baseline and then every six hours for the following 72 hours after randomization
  collected every 6 hours for 3 days
changes in the concentration of lactate(mmol/l) in the extracellular fluid of the skeletal muscle | Time Frame: At baseline and then every six hours for the following 72 hours after randomization
  collected every 6 hours for 3 days
changes in the concentration of pyruvate (µmol/l) in the extracellular fluid of the skeletal muscle | Time Frame: At baseline and then every six hours for the following 72 hours after randomization
  collected every 6 hours for 3 days
changes in the concentration of glycerol (µmol/l) in the extracellular fluid of the skeletal muscle | Time Frame: At baseline and then every six hours for the following 72 hours after randomization
  collected every 6 hours for 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Mustapha Ferjani, Study Director — Department of C ritical C are Medicine and Anesthesiology, Military Hospital of Tunis, Tunisia, Tunis, Tunisia
Locations (2):
- Tunisia (2):
  - Military hospital of tunis, Tunis, Mont Fleury
  - Military Hopital of Tunis, Tunis

IPD SHARING:
Plan to Share IPD: No